CLINICAL TRIAL: NCT06137794
Title: Application of the Anticoagulation Decision-making and Management Model Based on the "I-Anticoagulation" Tool in Patients With Atrial Fibrillation: A Prospective, Multicenter, Cluster Randomized Controlled Study
Brief Title: Application of "I-Anticoagulation"in Patients With Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIT-2023-0207
Record Dates: First submitted 2023-09-22; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation; Anticoagulants
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDM group (Experimental): The anticoagulation therapy of AF patients will be determined by clinicians with the use of "I-Anticoagulation", and AF patients will be managed using "I-Anticoagulation" during their anticoagulation therapy.
  Interventions: Other: Use of "I-Anticoagulation" to make the decision and manage patients
- Control group (No Intervention): AF patients in the control group will receive standard care.

INTERVENTIONS:
Other: Use of "I-Anticoagulation" to make the decision and manage patients — I-Anticoagulation will offer a flexible and efficient communication platform for healthcare professionals and AF patients. The tool is composed of two modules: an anticoagulation decision support system and a full-process patient management system.
  Arms: SDM group

SUMMARY:
The goal of this prospective, multicenter, cluster randomized controlled trial is to assess the effectiveness of a shared decision-making tool, "I-Anticoagulation", for anticoagulation management in AF patients. The main questions it aims to answer are:

* whether "I-Anticoagulation" could help improve the rational use of anticoagulants in AF patients;
* whether "I-Anticoagulation" could help increase the adherence and satisfaction of AF patients receiving anticoagulants.

The anticoagulation therapy of AF patients will be determined by clinicians with the use of "I-Anticoagulation", and AF patients will be managed using "I-Anticoagulation" during their anticoagulation therapy.

Researchers will compare the outcomes with the control group, in which patients with AF will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* patients who are 18 years or older and have received a new diagnosis of paroxysmal, persistent, or permanent AF confirmed by electrocardiogram (ECG) or 24-hour Holter monitors
* must be willing to participate in the study and sign the informed consent

Exclusion Criteria:

* those who are pregnant
* those whohave experienced therapeutic or subtherapeutic bleeding complications in the last 6 months
* those who have severe renal insufficiency (creatinine clearance rate, CrCl ≤ 20 ml/min)
* those who have severe hepatic insufficiency (Child-Pugh ≥ 10 points)
* those who have severe heart failure (cardiac function New York Heart Association, NYHA grade IV and above)
* those who have severe infection and respiratory failure
* those who are unable to comply with the study requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Any bleeding events | 1st, 3rd, 6th, 9th, and 12th months
  Any bleeding events, including both major and minor bleeding events. Major bleeding events include fatal haemorrhage, life-threatening bleeding, and severe bleeding requiring treatment or assessment. Severe bleeding can manifest as gastric intestinal haemorrhage, joint haematoma, retroperitoneal haemorrhage, fundus haemorrhage, urine, haemoptysis, or require blood transfusion of at least two units. Minor bleeding events, such as mild nasal hemorrhage, endoscopic haematuria, skin stasis, or mild hemorrhoids, do not lead to serious consequences.

SECONDARY OUTCOMES:
The accordance of stroke prophylaxis for AF according to current guidelines | 1st, 3rd, 6th, 9th, and 12th months
  The accordance of stroke prophylaxis for AF according to current guidelines, i.e., whether the prescriptions meet the recommendations on clinical guidelines, including the choice, usage and dosage of oral anticoagulants.
The percentage of time in the target INR range for patients using warfarin | 1st, 3rd, 6th, 9th, and 12th months
  The percentage of time in which the INR remains in the 1.8 to 3.0 target range across time for patients using warfarin.
The occurrences of major bleeding and thrombosis events | 1st, 3rd, 6th, 9th, and 12th months
  The occurrences of major bleeding and thrombosis events. Major bleeding events include fatal haemorrhage, life-threatening bleeding, and severe bleeding requiring treatment or assessment. Severe bleeding can manifest as gastric intestinal haemorrhage, joint haematoma, retroperitoneal haemorrhage, fundus haemorrhage, urine, haemoptysis, or require blood transfusion of at least two units. Thrombosis events, including ischaemic stroke, systemic embolism, and transient ischaemic attacks, will be confirmed by imaging methods such as ultrasound, CT, or MRI.
OAC knowledge of AF patients receiving anticoagulation therapy | 1st, 3rd, 6th, 9th, and 12th months
  The AKT comprises 28 items assessing general anticoagulation knowledge for all available OAC and a specific section for VKAs therapy.
OAC adherence of AF patients receiving anticoagulation therapy | 1st, 3rd, 6th, 9th, and 12th months
  The MARS-5 assesses common patterns of nonadherent behavior.
Satisfaction of AF patients receiving anticoagulation therapy | 1st, 3rd, 6th, 9th, and 12th months
  The ACTS evaluates the burdens and benefits of anticoagulation treatment and its overall impact.

IPD SHARING:
Plan to Share IPD: No